CLINICAL TRIAL: NCT05059665
Title: Specimen Collection for Multi-Analyte Blood-Test for Hepatocellular Carcinoma
Brief Title: Performance Evaluation (Sensitivity/Specificity) of HelioLiver Test for Detection of HCC
Acronym: ENCORE
Status: Completed | Type: Observational
Sponsor: Helio Genomics (Industry)
Collaborators: Laboratory for Advanced Medicine, Guangzhou (Unknown); Helio Health Inc., Irvine, CA (Unknown)
Responsible Party: Sponsor
Other Study IDs: LAM-2020-001
Record Dates: First submitted 2021-09-10; First posted 2021-09-28 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Hepatocellular Carcinoma by AJCC Stage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC Subjects: All subjects will be recently diagnosed with hepatocellular carcinoma as defined by at least one of the following criteria:
  * Subject has a ≥1 cm lesion exhibiting arterial phase hyperenhancement in combination with washout appearance by MRI and/or CT.
  * Subject has a lesion of any size indicated to be HCC due to capsule appearance by 4 phase CT scan and/or multiphase contrast enhanced MRI.
  * Subjects with a suspicious lesion of less than 2 cm must have HCC confirmed by both MRI and CT.
  * Subject has a biopsy that is positive for HCC.
  * Diagnostic imaging by multiphasic MRI or CT indicates a suspicious lesion on the liver, which is subsequently confirmed to be HCC by another method (biopsy, or surgical pathology).
  Interventions: Diagnostic Test: Helio Liver Test
- Surveillance Subjects: At-risk subjects with chronic liver disease undergoing routine imaging surveillance for HCC.
  Interventions: Diagnostic Test: Helio Liver Test

INTERVENTIONS:
Diagnostic Test: Helio Liver Test — De-identified whole blood and serum samples are collected for the purpose of evaluating the performance (sensitivity/specificity) of the HelioLiver Test for the detection of hepatocellular carcinoma (HCC).

SUMMARY:
De-identified whole blood and serum samples are collected for the purpose of evaluating the performance (sensitivity/specificity) of the HelioLiver Test for the detection of hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The purpose of this study is to define the performance characteristics (sensitivity and specificity) of the Helio Liver Test within a study population of subjects that have been diagnosed with liver cancer at various stages (I to IV) and for control subjects who have been confirmed to not have liver cancer by at least one imaging technique, such as ultrasound, MRI or CT. Control subjects will include patients who are at high-risk for liver cancer and have been recommended to undergo liver cancer surveillance, as well as patients who have non-HCC cancers to determine analytical specificity.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and Older (Adult, Older Adult)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who have been clinically diagnosed with HCC, or are negative for HCC after regular surveillance, or have been clinically diagnosed with non-HCC cancers will be enrolled. Approximately 500 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance (sensitivity/specificity) of the HelioLiver Test for early stage HCCs (Stage I and II) | 15 months
  performance evaluation (early stage, Stage I and II)
Evaluate the performance (sensitivity/specificity) of the HelioLiver Test for all stage HCCs | 15 months
  performance evaluation at all stages (I through IV)

CONTACTS AND LOCATIONS:
Overall Officials: RIchard Van Etten, MD, PhD, Principal Investigator — University of California, Irvine
Locations (2):
- China (2):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No